CLINICAL TRIAL: NCT06174428
Title: Validity of Viome's Oral/throat Cancer Test Among Patients with a Suspicion of Cancer
Brief Title: Validity of Viome's Oral/throat Cancer Test
Status: Recruiting | Type: Observational
Sponsor: Viome (Industry)
Responsible Party: Sponsor
Other Study IDs: V303
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Oral and Throat Cancer; Oropharyngeal Squamous Cell Carcinoma; Oral Squamous Cell Carcinoma
Keywords: OSCC; OPSCC; Oral Cancer; Throat cancer; Oral and Throat cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Mouth Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The Oral/Throat cancer test is intended for the qualitative detection of molecular features (human genes, microbial species and functions) associated with OSCC or OPSCC in saliva samples from adults with a suspicion of cancer. The system consists of the Saliva Collection and Transport Kit, the Viome laboratory process for metatranscriptomics, and the Viome analytical software that detects an RNA expression signature within a saliva sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Oral Squamous Cell Carcinoma (OSCC): OSCC case cohort will consist of patients with Oral Squamous Cell Carcinoma (all stages, locations), recruited from either primary or secondary care.
  Interventions: Device: Oral/Throat cancer test
- Oropharyngeal Squamous Cell Carcinoma (OPSCC): OPSCC case cohort will consist of patients with Oral Squamous Cell Carcinoma (all stages, locations), recruited from either primary or secondary care.
  Interventions: Device: Oral/Throat cancer test
- Cancer-free: Participants will be recruited following clinical adjudication with self-reported confirmation of no cancer and from primary and secondary care facilities.
  Interventions: Device: Oral/Throat cancer test

INTERVENTIONS:
Device: Oral/Throat cancer test — The Oral/Throat cancer test is intended for the qualitative detection of molecular features (human genes, microbial species and functions) associated with Oral Squamous Cell Carcinoma (OSCC) or OroPharyngeal Squamous Cell Carcinoma (OPSCC) in saliva samples from adults with a suspicion of cancer. A positive result from CDOT may indicate the presence of OSCC or OPSCC. The device is intended as a diagnostic aid for clinicians when assessing patients with suspected OSCC or OPSCC who may benefit from follow-up diagnosis and treatment. The device is not intended for a definitive diagnosis.

SUMMARY:
A total of at least 1,000 participants with suspicion of cancer including at least 107 subjects who will be diagnosed with OSCC or OPSCC will be enrolled from either primary or secondary care centers in the U.S. Clinicians will use Viome collection kits to collect saliva samples from eligible patients.

DETAILED DESCRIPTION:
This is a prospective, multi-center study. Subjects with OSCC or OPSCC will be enrolled from four primary and secondary care centers in the U.S. Study samples will be collected by the clinicians at the study sites using Viome saliva sample collection kits. Patients will continue with their current health plan and confirm diagnosis following the standard of care of surgical biopsy with histology if needed. If a biopsy is performed, the result of the biopsy will be compared with the result of the Viome kit. If no biopsy is performed, the Viome test result will be compared with the physician's assessment based on clinical judgment. Patients with a positive result from histology will not receive the results of the Viome kit, and it will not play any part in the clinical management of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent prior to any study-specific procedures are performed
* Willing and able to follow the study instructions, as described in the recruitment letter
* Adults (18 years old or older)
* Suspicion of OSCC or OPSCC on clinical presentation by a clinician

Exclusion Criteria:

* Pregnancy
* Use of fertility enhancing medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will comprise patients who attend (1) a primary care center (typically dentist offices) and are identified with a suspicion of cancer based on a clinical presentation or (2) a secondary care center (typically hospitals) following the finding of a suspicious lesion or symptom. Secondary care centers include clinical sites where specialists such as oncologists or oral and maxillofacial surgeons (also called head and neck surgeons) perform visual and tactile oral examinations and biopsies to detect oral cancer. They are also known as ear, nose, and throat (ENT) doctors or otolaryngologists.
  Women or minorities are not excluded from this study. In order to calculate an estimated number of samples in each demographic category we performed stratified random sampling. We used the SEER Program to calculate oral and throat cancer prevalence for each of the demographic categories.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | Through study completion, an average of 18 months
  Oral/Throat cancer test's ability to designate an individual with disease as positive
Specificity | Through study completion, an average of 18 months
  Oral/Throat cancer test's ability to designate an individual who does not have a disease as negative
Positive Post Test Probability (PPV) | Through study completion, an average of 18 months
  The probability of having the target condition if the test falls out positive
Negative Post Test Probability (NPV) | Through study completion, an average of 18 months
  The probability of having the target condition if the test falls out negative

SECONDARY OUTCOMES:
Sensitivity by care center (primary and secondary) | Through study completion, an average of 18 months
  Oral/Throat cancer test's ability to designate an individual with disease as positive
Sensitivity by age | Through study completion, an average of 18 months
  Oral/Throat cancer test's ability to designate an individual with disease as positive
Sensitivity by sex | Through study completion, an average of 18 months
  Oral/Throat cancer test's ability to designate an individual with disease as positive
Sensitivity by race | Through study completion, an average of 18 months
  Oral/Throat cancer test's ability to designate an individual with disease as positive
Sensitivity by smoking history | Through study completion, an average of 18 months
  Oral/Throat cancer test's ability to designate an individual with disease as positive
Sensitivity by oral cancer type (OSCC or OPSCC) | Through study completion, an average of 18 months
  One measure post treatment
Sensitivity by disease stage (I, II, III, and IV) | Through study completion, an average of 18 months
  Oral/Throat cancer test's ability to designate an individual with disease as positive
Sensitivity by metastasis | Through study completion, an average of 18 months
  Oral/Throat cancer test's ability to designate an individual with disease as positive
Sensitivity by HPV status | Through study completion, an average of 18 months
  Oral/Throat cancer test's ability to designate an individual with disease as positive
Sensitivity by recurrent cancer | Through study completion, an average of 18 months
  Oral/Throat cancer test's ability to designate an individual with disease as positive
Specificity by care center (primary and secondary) | Through study completion, an average of 18 months
  One measure post treatment
Specificity by age | Through study completion, an average of 18 months
  Oral/Throat cancer test's ability to designate an individual who does not have a disease as negative
Specificity by sex | Through study completion, an average of 18 months
  Oral/Throat cancer test's ability to designate an individual who does not have a disease as negative
Specificity by race | Through study completion, an average of 18 months
  Oral/Throat cancer test's ability to designate an individual who does not have a disease as negative
Specificity by smoking history | Through study completion, an average of 18 months
  Oral/Throat cancer test's ability to designate an individual who does not have a disease as negative
Specificity by oral cancer type (OSCC or OPSCC) | Through study completion, an average of 18 months
  Oral/Throat cancer test's ability to designate an individual who does not have a disease as negative
Specificity by disease stage (I, II, III, and IV) | Through study completion, an average of 18 months
  Oral/Throat cancer test's ability to designate an individual who does not have a disease as negative
Specificity by metastasis | Through study completion, an average of 18 months
  Oral/Throat cancer test's ability to designate an individual who does not have a disease as negative
Specificity by HPV status | Through study completion, an average of 18 months
  Oral/Throat cancer test's ability to designate an individual who does not have a disease as negative
Specificity by recurrent cancer | Through study completion, an average of 18 months
  Oral/Throat cancer test's ability to designate an individual who does not have a disease as negative

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Julian, Principal Investigator — Viome
Locations (2):
- United States (2):
  - Missouri School of Dentistry & Oral Health, St Louis, Missouri
  - UTHSC, Memphis, Tennessee